CLINICAL TRIAL: NCT03156998
Title: Patients' Compliance to Home Nebulizer Therapy for Children's Asthma in China An Observational Study to Investigate the Compliance of Home Nebulizer Therapy Among Children Aged 0-14 Years Old Clinically Diagnosed With Asthma
Brief Title: Patients' Compliance to Home Nebulizer Therapy for Children's Asthma in China
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5252R00001
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Paediatric Asthma
Keywords: CARE; Paediatric asthma; Compliance; Home nebulizer
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study to investigate the compliance of home nebulizer therapy among children aged 0-14 years old clinically diagnosed with asthma

DETAILED DESCRIPTION:
Asthma is the most common chronic disease of childhood and the leading causes of childhood morbidity from chronic disease (GINA 2016). It is clear that inhaled corticosteroid (ICS) is foundation of asthma treatment and recommended both in Global Initiative for Asthma (GINA) and Chinese paediatric asthma diagnosis and treatment guideline. But the well-controlled rate of asthma was not ideal. National Parents of Asthmatic Children KAP Project Team (China) showed that 66.0% asthmatic children had asthma attacks in the past 12 months, 26.8% asthmatic children had visited the emergency department and 16.2% asthmatic children had been hospitalized. (Asthmatic Children KAP project team, 2013) .A few studies showed an increased risk of uncontrolled asthma or an asthma exacerbation in children with lower compliance (Jentzsch NS, 2012; Milgrom H, 1996). Poor compliance to inhaled corticosteroids may also contribute to poor asthma control level and asthma mortality (GINA 2016). Home nebulizer therapy has been recommended in GINA and Chinese Paediatric asthma diagnosis and treatment guideline. Compare to other inhalers, delivering ICS through nebulizer therapy need minimal patient's cooperation and normal breathing pattern (Deborah Elliott, 2011), but there are no studies to show the compliance of home nebulizer therapy in Chinese clinical practice. So we aim to investigate the compliance to home nebulizer therapy, and try to explore the related risk factor with poor compliance in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 0-14 years old, clinical diagnosed as asthma according to Chinese paediatric asthma diagnosis and treatment guideline
2. Prescribed home nebulizer therapy for at least 3 month
3. The guardians must sign the Informed Consent Form; Subjects who can make decision by him/herself must also sign the Informed Consent Form

Diagnosis of paediatric asthma:

The patient who fulfil criteria 1 to 4 or criteria 4 plus any item of criteria 5 could be diagnosed as paediatric asthma.

1. Recurrent respiratory symptoms (wheeze, cough, dyspnoea, chest tightness), typically worse at night/early morning, exacerbated by exercise, viral infection, smoke, dust, pets, mold, dampness, weather changes, laughing, crying, allergens.
2. A musical, high-pitched whistling sound could be detected in both sides of the lung by auscultation of the chest. The wheezing is usually during exhalation.
3. Symptoms/signs above could be relieved automatically or by anti-asthmatic treatment.
4. Exclusion of the other diseases, which also could cause wheeze, cough, dyspnoea, chest tightness.
5. Atypical symptoms/signs without any wheeze or whistling sound (at least fulfil one of the following criteria):

1) The results of bronchial provocation test is positive. 2) Demonstrating reversible airflow limitation: i. The result of bronchial dilation test is positive. ii. Anti-asthmatic treatment is effective for lung function improvement. 3) The ratio of daily variation of PEF (consecutively more than two weeks) is more than 13%.

Exclusion Criteria:

1. Allergy to any inhaler cortical steroid
2. Presenting with differential diagnosis of asthma such as congenital heart disease, gastro-oesophageal reflux, bronchopulmonary dysplasis, bronchiolitis obliterans, etc
3. Parents/Guardian have problem in expression, understanding, writing and reading in Chinese judged by the investigator
4. Subjects are participating other on-going clinical studies
5. Subjects with other diseases that may interfere the study results judged by the investigators

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 500 children aged 0-14 years old who are diagnosed with asthma and prescribed home nebulizer therapy treatment at tier-3 hospitals by investigators according to Chinese paediatric asthma diagnosis and treatment guideline
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Median treatment compliance (%) derived using actual treatment frequency (monitored by electronic chips) divided by prescribed frequency | From 3 June 2017 to 3 March 2018, an expected average of 3 months

SECONDARY OUTCOMES:
Proportion of patients in different treatment compliance levels (<50%, 50 %≤-< 80%, 80%≤-≤120%, >120%) monitored by electric chips | From 3 June 2017 to 3 March 2018, an expected average of 3 months
Median treatment compliance (%) reported by caregivers derived using actual doses divided by prescribed doses | From 3 June 2017 to 3 March 2018, an expected average of 3 months
Proportion of patients in difference compliance levels reported by caregivers | From 3 June 2017 to 3 March 2018, an expected average of 3 months
Proportion of patients by severity | From 3 June 2017 to 3 March 2018, an expected average of 3 months
Factors associated with treatment compliance | From 3 June 2017 to 3 March 2018, an expected average of 3 months
The proportion of asthma control status (controlled, partly controlled and uncontrolled asthma) according to GINA 2016 definition at visit 2 to 4 overall and by compliance level. | From 3 June 2017 to 3 March 2018, an expected average of 3 months
The proportion of asthma control status according to TRACK for subjects under 5 years old | From 3 June 2017 to 3 March 2018, an expected average of 3 months
Factors associated with control levels (controlled, partly controlled and uncontrolled asthma) | From 3 June 2017 to 3 March 2018, an expected average of 3 months

OTHER OUTCOMES:
Direct health expenditure of asthma treatment and management | From 3 June 2017 to 3 March 2018, an expected average of 3 months
caregiver's loss of working days | From 3 June 2017 to 3 March 2018, an expected average of 3 months
children's loss of kindergarten/school days | From 3 June 2017 to 3 March 2018, an expected average of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Deyu Zhao, Principal Investigator — Nanjing Children's Hospital
Locations (12):
- China (12):
  - Facility, Bengbu, Anhui
  - Facility, Hefei, Anhui
  - Facility, Lanzhou, Gansu
  - Facility, Guangzhou, Guangdong
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Facility, Nanjing, Jiangsu
  - Facility, Wuxi, Jiangsu
  - Facility, Xuzhou, Jiangsu
  - Facility, Nanchang, Jiangxi
  - Facility, Shenyang, Liaoning
  - Facility, Chengdu, Sichuan
  - Facility, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao D, Chen D, Li L, Zou Y, Shang Y, Zhang C, Zhang L, Pan J, Chen Q, Ai T, Ni Q. CARE: an observational study of adherence to home nebulizer therapy among children with asthma. Ther Adv Respir Dis. 2021 Jan-Dec;15:1753466620986391. doi: 10.1177/1753466620986391. PMID 33541235
- See also: CSR synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14693&filename=CARE_study_(D5252R00001)_CSR_synopsis.pdf